CLINICAL TRIAL: NCT01131416
Title: The Effects of Gum Chewing on Bowel Function Recovery Following Cesarean Section: Randomized Controlled Trial
Brief Title: The Effects of Gum Chewing on Bowel Function Recovery Following Cesarean Section
Acronym: GUM01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Kittipat Charoenkwan, M.D., Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10FEB010938
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Paralytic Ileus
MeSH Terms: conditions — Intestinal Pseudo-Obstruction | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gum chewing (Experimental): Gum chewing (30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in addition to conventional postoperative feeding schedule
  Interventions: Behavioral: Gum chewing
- Conventional (No Intervention): Conventional postoperative feeding schedule

INTERVENTIONS:
Behavioral: Gum chewing — Gum chewing (30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in addition to conventional postoperative feeding schedule
  Arms: Gum chewing

SUMMARY:
Following all abdominal surgery, paralytic ileus commonly develops. Surgeons have traditionally withheld postoperative oral intake until the return of bowel function to prevent related complications. Gum chewing can stimulates bowel movement and promotes the return of bowel function through the cephalic-vagal reflex and increased intestinal enzymes secretion.

The objectives of this study are to examine effects of adding gum chewing to the conventional postoperative feeding regimen on the return of bowel function, its related complications, and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing cesarean delivery

Exclusion Criteria:

* Perioperative hyperalimentation
* Recent chemotherapy
* Concurrent bowel surgery
* Previous bowel surgery
* Concurrent bowel obstruction
* History of inflammatory bowel diseases
* Previous abdominal/pelvic radiation
* Postoperative placement of endotracheal tube/nasogastric tube
* Postoperative admission to intensive care unit

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Postoperative interval until the first flatus | Up to 7 days after delivery

SECONDARY OUTCOMES:
Postoperative interval until the first passage of stool | Up to 7 days after delivery
Clinically significant postoperative ileus | Up to 7 days after delivery
Postoperative hospital stay | Up to 7 days after delivery
Related complications | Up to 7 days after delivery
Patients' satisfaction | Up to 7 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand